CLINICAL TRIAL: NCT00179452
Title: Is Yoga Safe for Patients With Epilepsy?
Brief Title: Yoga for Patients With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Kaarkuzhali Babu Krishnamurthy, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2003P000337
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: epilepsy, yoga
MeSH Terms: conditions — Epilepsy | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Subjects invited to participate in yoga practice.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga

SUMMARY:
To establish the safety and feasibility of having patients with epilepsy perform yoga.

DETAILED DESCRIPTION:
Subjects will keep logs of seizure frequency prior to, during, and following training in a yoga regimen. Instruction in the yoga regimen will occur at BIDMC, and home practice following classroom instruction will occur as part of the study. Side effects, changes in seizure frequency, and quality of life assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to give full informed consent.
2. Must have one or more of the following seizure types: simple partial, complex partial, or secondarily generalized.
3. Age 18-64.
4. Must have 4-20 during the baseline phase.
5. Must have medical clearance from their primary care giver sufficient to allow for participation in yoga exercises.
6. Must be stable enough to allow for all anticonvulsant levels to remain constant for the duration of the study.

Exclusion Criteria:

1. Having primary generalized epilepsy or atonic seizures.
2. Having a history of status epilepticus in the past two years.
3. Any medical problem that would preclude participation in a yoga class.
4. Nonepileptic or psychogenic seizures.
5. Pregnancy.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of life assessments. | 3 months
Improvement in mood. | 3 months

SECONDARY OUTCOMES:
Improvement in seizure control. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kaarkuzhali Krishanmurthy, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share as was not included in original protocol as approved by the IRB, so subject consent was not obtained.